CLINICAL TRIAL: NCT01091480
Title: French Hypertrophic Cardiomyopathy Observatory
Acronym: REMY
Status: Recruiting | Type: Observational
Sponsor: French Cardiology Society (Other)
Responsible Party: Principal Investigator, Hagege Albert, Professor, French Cardiology Society
Other Study IDs: 09273
Record Dates: First submitted 2010-03-08; First posted 2010-03-24 (Estimated); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Hypertrophic Cardiomyopathy
Keywords: Hypertrophic cardiomyopathy; Observatory; LVH
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Systematic search for predisposition genes and Fabry disease in patients with hypertrophic cardiomyopathy (GE-REMY) with blood sampling at baseline or during a consultation normally scheduled as part of the management of this pathology
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with HCM: Patients ≥ 15 years with HCM(sarcomere of origin or not) defined by an ultrasound thickness of the left ventricle ≥ 13 mm if familial or ≥ 15 mm if sporadic

SUMMARY:
Hypertrophic cardiomyopathy (Hypertrophic CardioMyopathy=HCM) remains a poorly understood disease with an assumption insufficiently codified. There is no data available in France on the profile of patients, diagnostic methods and assessment and therapeutic use.

The purpose of this study is to establish a monitoring of patients with HCM (sarcomere of origin or not) in France (diagnosis, treatment)

DETAILED DESCRIPTION:
This both retrospective and prospective study is proposed to cardiology services 50 hospitals in France. A cardiologist referral is designated for each facility.

The following data will be collected by the physician during the initial hospitalization

* Demographics
* Geographic origin of patient
* Clinical data: criteria for inclusion and non-inclusion data HCM general, Doppler ultrasound, personal history, family history
* Reviews made: non-organic, biological
* Family Survey,
* Treatments: Medical, Electrical, invasive
* Data from hospital

The follow-up to 18 months, 3 years and 5 years will be conducted by clinical-research-technicians of the French Society of Cardiology, an application will be made to municipalities of birth and mail a letter to physicians and patients.

The following data will be collected:

* Vital status
* Data from hospital
* Reviews made: non-organic, biological
* Treatments: Medical, Electrical, invasive

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 15 years old
* Patient with HCM defined by an ultrasound thickness of the left ventricle ≥ 13 mm if familial or ≥ 15 mm if sporadic

Exclusion Criteria:

* Expressed refusal to participate in the study
* Significant aortic stenosis (<1 cm ²)

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients ≥ 15 years old with HCM (sarcomere of origin or not) defined by an ultrasound thickness of the left ventricle ≥ 13 mm if familial or ≥ 15 mm if sporadic
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2010-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Event-free survival | 3 years

SECONDARY OUTCOMES:
Diagnostic methods | 0 day
  Define the profile of patients with HCM in France, diagnostic methods, evaluation (diagnostic investigation and family) and therapeutic. Who are the patients CMH France? (rules discovery, clinical presentation) and how are assumed the HCM in France? (examinations, hospitalizations, treatments, procedures for the family survey).

CONTACTS AND LOCATIONS:
Locations (1):
- European Georges Pompidou Hospital, Paris, France

REFERENCES:
- [Result] Mirabel M, Damy T, Donal E, Huttin O, Labombarda F, Eicher JC, Cervino C, Laurito M, Offredo L, Tafflet M, Jouven X, Giura G, Desnos M, Jeunemaitre X, Empana JP, Charron P, Habib G, Reant P, Hagege A; REMY working group of the French Society of Cardiology. Influence of centre expertise on the diagnosis and management of hypertrophic cardiomyopathy: A study from the French register of hypertrophic cardiomyopathy (REMY). Int J Cardiol. 2019 Jan 15;275:107-113. doi: 10.1016/j.ijcard.2018.09.083. Epub 2018 Sep 28. PMID 30316646
- [Derived] Sakhi H, Soulat G, Craiem D, Gencer U, Lamy J, Stipechi V, Puscas T, Hulot JS, Hagege A, Mousseaux E. Association of Impaired Left Ventricular Mitral Filling from 4D Flow Cardiac MRI and Prognosis of Hypertrophic Cardiomyopathy. Radiol Cardiothorac Imaging. 2024 Apr;6(2):e230198. doi: 10.1148/ryct.230198. PMID 38512023